CLINICAL TRIAL: NCT05903040
Title: Effectiveness and Tolerability of Lasmiditan as Acute Migraine Treatment: a Prospective, Multicentric, Cohort Study
Brief Title: Ditan Acute tReatments: Effectiveness and Tolerability (DART)
Acronym: DART
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Società Italiana per lo Studio delle Cefalee (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Università degli Studi dell'Aquila (Other); University of Roma La Sapienza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Ospedale di Piove di Sacco (Unknown); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); A.O.U. Città della Salute e della Scienza (Other); Cliniche Humanitas Gavazzeni (Other); University of Campania Luigi Vanvitelli (Other); Ospedale Santo Stefano (Other); Azienda Policlinico Umberto I (Other); Auxologico San Luca (Other); Asst Degli Spedali Civili Di Brescia (Other); Carlo Besta Neurological Institute (Other)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher, University of Modena and Reggio Emilia
Other Study IDs: RICe_2
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: Headache; Medication overuse headache; Pain; Ditan; Triptan
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache; Headache Disorders, Secondary; Pain | interventions — lasmiditan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by an episodic pattern (< 15 monthly headache days) migraine with or without aura according to ICHD-III criteria.
  Interventions: Drug: Lasmiditan
- Chronic migraine: Patients affected by chronic migraine according to ICHD-III criteria.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Patients using Lasmiditan 50-100-200 mg oral tablet to treat acute migraine attacks

SUMMARY:
The purpose of this prospective and multicentric study is to evaluate the effectiveness and tolerability of lasmiditan as acute migraine treatment in a cohort of episodic or chronic migraine patients.

DETAILED DESCRIPTION:
Lasmiditan is a serotonin 5-HT1F receptor agonist. It is available in three different dosages (namely 50, 100 and 200 mg) with oral administration. Phase 3 double-blind randomized controlled studies demonstrated its effectiveness 2h post-dose in a single migraine attack and consistent effectiveness across four different attacks.

The lack of vasoconstrictive activity allow its use also in patients with cardiovascular medical history. This finding was also confirmed in a real-world study. As it is a small molecule with access to the central nervous system predominant adverse events are CNS-related (as dizziness, somnolence and paraesthesia).

In this prospective multicentric study the Investigators aim to evaluate lasmiditan effectiveness and tolerability as acute migraine treatment in a real-world setting. Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline demographic and clinical data will be collected at the baseline. Patients will be asked to treat their next migraine attack with lasmiditan 50 - 100 - 200 mg oral tablet.

Data will be collected at baseline, during at least 4 migraine attacks treated with lasmiditan and at 3 months follow-up.

Subjects will be asked to complete assessment of their migraine attack at baseline and at 30 - 60 - 90 and 120 minutes after administration of the acute treatment for at least four migraine attacks. A final timepoint at 24 hours post-dose will be assessed only for the first attack.

Data collection will focus on: i) demographic data, ii) migraine history, iii) pain level and evolution, iv) presence and evolution of migraine associated symptoms, most bothersome symptom and aura, v) migraine associated disability, vi) patients's global impression of change (PGIC) and evaluation on the acute treatment (Migraine-ACT), vii) tolerability and eventual treatment-emergent adverse events. The online database REDCap will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III).

At least 3 MMDs

* Good compliance to study procedures
* Availability of headache diary at least of the preceding months before enrollment

Exclusion Criteria:

* Subjects with contraindications for use of ditans;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion might interfere with study assessments;
* medical comorbidities that could interfere with study results;
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for lasmiditan use for acute migraine treatments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Headache pain freedom at 2 hours post dose during the first attack | 2 hours post-dose
  The percentage of subjects that report no headache pain at 2 hours after drug intake. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Occurrence of treatment-emergent adverse events | 12 weeks
  To evaluate the safety and tolerability of Lasmiditan in migraine subjects

SECONDARY OUTCOMES:
Headache pain freedom at 2 hours post dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that report no headache pain at 2 hours after drug intake across all' treated attacks. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache pain relief at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that report mild or none headache pain at 2 hours after drug intake during the first attack. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache pain relief at 2 hours post-dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that report mild or none headache pain at 2 hours after drug intake across all treated attack. Pain will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Ability to function normally at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that self-report no functional disability at 2 hours post-dose. Functional disability will be assessed through the Functional Disability Scale (FDS), a four-point scale: normal, mildly impaired, severely impaired, requires daily activities interruption.
Ability to function normally at 2 hours post-dose across all treated attacks | 2 hours post-dose for all treated attacks
  The percentage of subjects that self-report no functional disability at 2 hours post-dose. Functional disability will be assessed through the Functional Disability Scale (FDS), a four-point scale: normal, mildly impaired, severely impaired, requires daily activities interruption.
Freedom from the most bothersome symptom (MBS) associated with migraine at 2 hours post-dose during the first attack | 2 hours post-dose
  The percentage of subjects that report complete MBS resolution at 2 hours after drug intake. MBS will be measured on a 4 point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).
Headache recurrence for the first-attack | between 2 hours and 24 hours post-dose
  Percentage of subjects who became pain free at 2 hours post-dose and report new headache pain within 24 hours post-dose.
Rescue medications use for the first attack | between 2 hours and 24 hours post dose
  Percentage of subjects who take a rescue medication after 2 hour post-dose. Rescue medications will be measured using a binary scale (0=no consumption, 1=consumption)
Treatment satisfaction | 2 hours post-dose for all treated attacks
  Level of patients' self-reported satisfaction which will be measured on a 0-10 visual analogue scale (0=no satisfaction, 10= the highest satisfaction) and Patients Global Impression of Change (0= no changing, 7= a change that makes the difference).
Self-reported treatment effectiveness | 12 weeks
  Level of patients' self-reported treatment effectiveness measured by Migraine Assessment of Current Therapy (migraine ACT) a 4-item questionnaire about treatment effectiveness and daily life repercussions.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ashina M, Reuter U, Smith T, Krikke-Workel J, Klise SR, Bragg S, Doty EG, Dowsett SA, Lin Q, Krege JH. Randomized, controlled trial of lasmiditan over four migraine attacks: Findings from the CENTURION study. Cephalalgia. 2021 Mar;41(3):294-304. doi: 10.1177/0333102421989232. Epub 2021 Feb 4. PMID 33541117
- [Background] Goadsby PJ, Wietecha LA, Dennehy EB, Kuca B, Case MG, Aurora SK, Gaul C. Phase 3 randomized, placebo-controlled, double-blind study of lasmiditan for acute treatment of migraine. Brain. 2019 Jul 1;142(7):1894-1904. doi: 10.1093/brain/awz134. PMID 31132795
- [Derived] Vaghi G, Iannone LF, Corrado M, De Santis F, Romozzi M, Sebastianelli G, Dalla Volta G, Bolchini M, Burgalassi A, De Cesaris F, Albanese M, Mercuri Biagio N, Ornello R, Sacco S, Pistoia F, Saporito G, Casillo F, Avino G, Granato A, Russo A, Silvestro M, Vollono C, Trimboli M, Doretti A, Valente M, Cevoli S, Mampreso E, Tassorelli C, De Icco R. Effectiveness and tolerability of lasmiditan in the acute treatment of migraine: a real-world, prospective, multicentric study (DART study). Ther Adv Neurol Disord. 2025 Dec 21;18:17562864251381886. doi: 10.1177/17562864251381886. eCollection 2025. PMID 41446321